## **Protocol Changes**

Changes made from version 2 (published May 14, 2019) to version 3 (December 3, 2020)

- Two new investigators added (title page):
  - Mads Tofte Gregers, Copenhagen Emergency Medical Services, Ballerup, Denmark Annette Kjær Ersbøll, National Institute of Public Health, University of Southern Denmark, Copenhagen, Denmark
  - One investigator removed (title page):
  - Lena Karlsson, Copenhagen Emergency Medical Services, Ballerup, Denmark
- Power calculation changed. Baseline survival is increased from 12% to 15% based on data from 2018 from the Danish Cardiac Arrest Registry that has been published recently. Effect estimate for stratum 1 has been decreased from 35% to 25%. The new power calculation, including these new data, results in a sample size of 536 patient for both stratum 1 and 2. Since we are expecting 64% to be true OHCA and a citizen responder only arriving before EMS in 40% of the cases, we will include 2094 patients in stratum 1 and 2094 patients in stratum 2 (section 5.2)
- Length of study changed from 4 years to up to 8 years, and total included patients changed to approximately 4200 because of changes in power calculation (multiple sections)
- New wording for the approval from the Ethics Committee and addition of add-on approvals
  from the Danish Patient Safety Authority for data collection in 2019 and 2020 (Scientific
  summary and section 8)
- Secondary outcome. Neurological intact survival will be assessed at hospital discharge through patient's charts, not at 30 days. This is changed in multiple sections and a new data source has been added to section 4.12
- Safety outcome. Psychological impact will not be assessed at 4 weeks but assessed through a survey sent out 90 minutes after activation. Non-responders will be followed-up by phone call, text message or e-mail.
- Stratum 3 will not be included in analyses since this stratum is assumed to be very small.
- One subgroup has been deleted (arrival of citizen responders prior to EMS, since this is not
  assessable for the control group). The subgroup assessing OHCAs in public and residential
  settings has been divided op into two separate groups.
- The wording *heart runner* has been changed to *citizen responder* throughout the protocol

• Corrections of grammar and minor typing errors throughout the protocol